CLINICAL TRIAL: NCT02199795
Title: Functional Electrical Stimulation Mediated Neuroplasticity: Lower Extremity CCNMES in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jayme Knutson, Assistant Professor, Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23HD060689 (NIH); K23HD060689 (NIH)
Record Dates: First submitted 2014-06-23; First posted 2014-07-24 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Stroke; Hemiparesis; Footdrop
Keywords: stroke; hemiplegia; footdrop; electrical stimulation
MeSH Terms: conditions — Stroke; Paresis; Peroneal Neuropathies; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- CCNMES (Experimental): Contralaterally Controlled Neuromuscular Electrical Stimulation (CCNMES): CCNMES uses electrical stimulation to move the weaker ankle up and down. The user will control the stimulation using the other (stronger) ankle. A special sock is worn on the stronger ankle. When the stronger ankle is moved, a signal is sent from a sensor on the sock to the electrical stimulator. The stimulator then sends stimulation to the weaker ankle which causes it to move. Sound and light cues coming from the stimulator will tell the user when to move the stronger ankle and when to relax.
  Interventions: Device: Contralaterally Controlled Neuromuscular Electrical Stimulation
- Cyclic NMES (Active Comparator): Cyclic Neuromuscular Electrical Stimulation (NMES) uses automatic, repetitive electrical stimulation to stimulate the muscles in order to move the weaker ankle up and down.
  Interventions: Device: Cyclic Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Contralaterally Controlled Neuromuscular Electrical Stimulation
  Arms: CCNMES
Device: Cyclic Neuromuscular Electrical Stimulation
  Arms: Cyclic NMES

SUMMARY:
This is a small pilot randomized controlled trial which will enroll both subacute (<6 mos) and chronic (>6 mos) stroke survivors with ankle dorsiflexion weakness. The subjects will be randomized to Contralaterally Controlled Neuromuscular Electrical Stimulation (CCNMES) versus control. The primary objective of this study is to compare the effect of 6-weeks of lower extremity CCNMES, applied in an anti-phase application, on motor impairment and functional mobility to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 75 years
* Minimum of 2 wks from a first clinical non-hemorrhagic or hemorrhagic stroke
* Medically stable
* Unilateral lower extremity hemiparesis
* Ankle dorsiflexor strength of ≤4/5 on the Medical Research Council scale, while seated
* NMES of the paretic ankle dorsiflexors produces ankle dorsiflexion to neutral without pain.
* Full voluntary ROM of the contralateral ankle
* Skin intact on bilateral lower extremities
* Able to don the NMES system or caregiver available to assist with device if needed.
* Able to hear and respond to stimulator auditory cues
* Able to follow 3-stage commands
* Able to recall 2 of 3 items after 30 minutes
* Cognition and communication adequate for safe use of the device based on neurological assessment by physician principal investigator

Exclusion Criteria:

* Severely impaired cognition and communication
* History of peroneal nerve injury
* History of Parkinson's, spinal cord injury, traumatic brain injury, or multiple sclerosis
* Uncontrolled seizure disorder
* Uncompensated hemi-neglect (extinguishing to double simultaneous stimulation)
* Edema of the paretic lower extremity
* Absent sensation of paretic lower extremity
* Evidence of deep venous thrombosis or thromboembolism
* History of cardiac arrhythmias with hemodynamic instability
* Cardiac pacemaker or other implanted electronic system
* Botulinum toxin injections to any lower extremity muscle in the last 3 months
* Pregnancy
* Symptomatic peripheral neuropathy
* Current use of psychoactive medications (except selective serotonin reuptake inhibitor and serotonin-norepinephrine reuptake inhibitor antidepressants)
* Acetylcholinesterase inhibitor usage
* Unstable asthmatic condition
* Metallic implants (including clips and/or wires)
* Prosthetic heart valves
* Cardiac, renal or other stent
* History of claustrophobia
* Low visual acuity
* Body weight or body habitus not compatible to MRI machine
* Medical, psychological, or social concern identified by the principal investigator or co-investigator which suggests inappropriateness of subject participation

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne R. Sheffler, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knutson JS, Hansen K, Nagy J, Bailey SN, Gunzler DD, Sheffler LR, Chae J. Contralaterally controlled neuromuscular electrical stimulation for recovery of ankle dorsiflexion: a pilot randomized controlled trial in patients with chronic post-stroke hemiplegia. Am J Phys Med Rehabil. 2013 Aug;92(8):656-65. doi: 10.1097/PHM.0b013e31829b4c16. PMID 23867888
- [Background] Knutson JS, Chae J. A novel neuromuscular electrical stimulation treatment for recovery of ankle dorsiflexion in chronic hemiplegia: a case series pilot study. Am J Phys Med Rehabil. 2010 Aug;89(8):672-82. doi: 10.1097/PHM.0b013e3181e29bd7. PMID 20531158
- [Background] Swinnen SP. Intermanual coordination: from behavioural principles to neural-network interactions. Nat Rev Neurosci. 2002 May;3(5):348-59. doi: 10.1038/nrn807. PMID 11988774
- [Background] Kawashima N, Nozaki D, Abe MO, Akai M, Nakazawa K. Alternate leg movement amplifies locomotor-like muscle activity in spinal cord injured persons. J Neurophysiol. 2005 Feb;93(2):777-85. doi: 10.1152/jn.00817.2004. Epub 2004 Sep 22. PMID 15385590
- [Background] Vasudevan EV, Zehr EP. Multi-frequency arm cycling reveals bilateral locomotor coupling to increase movement symmetry. Exp Brain Res. 2011 Jun;211(2):299-312. doi: 10.1007/s00221-011-2687-y. Epub 2011 Apr 23. PMID 21516330
- See also: Cleveland Functional Electrical Stimulation Center — http://fescenter.org/index.php

RESULTS

PARTICIPANT FLOW:
Groups:
- CCNMES: Contralaterally Controlled Neuromuscular Electrical Stimulation (CCNMES): CCNMES uses electrical stimulation to move the weaker ankle up and down. The user will control the stimulation using the other (stronger) ankle. A special sock is worn on the stronger ankle. When the stronger ankle is moved, a signal is sent from a sensor on the sock to the electrical stimulator. The stimulator then sends stimulation to the weaker ankle which causes it to move. Sound and light cues coming from the stimulator will tell the user when to move the stronger ankle and when to relax.
  Contralaterally Controlled Neuromuscular Electrical Stimulation
- Cyclic NMES: Cyclic Neuromuscular Electrical Stimulation (NMES) uses automatic, repetitive electrical stimulation to stimulate the muscles in order to move the weaker ankle up and down.
  Cyclic Neuromuscular Electrical Stimulation
Period: Overall Study
Arm/Group | CCNMES | Cyclic NMES
Started | 4 | 3
Completed | 2 | 3
Not Completed | 2 | 0
Not completed — no longer met inclusion criteria | 1 | 0
Not completed — withdrew due to shoulder pain | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCNMES | Cyclic NMES | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (7.1) | 57 (31.8) | 44.2 (28.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Lower Extremity Fugl-Meyer Score at End of Treatment
Description: The Lower Extremity Fugl-Meyer (LEFM) Assessment is a measure of lower limb motor impairment. Participants are asked to attempt to perform a list of isolated and simultaneous movements of the hip, knee, and ankle that take into account synergy patterns, isolated strength, coordination, and hypertonia. Each movement attempt is graded on a 3-point ordinal scale (0, cannot perform; 1, perform partially; and 2, perform fully) and these subscores are summed to provide a maximum score of 34, minimum score of 0 (i.e., full scale range 0-34).
  Higher scores are considered to be a better outcome. For each individual, the score prior to treatment was subtracted from the score at end of the 6-week treatment. Then for each treatment group, these change scores were averaged.
Time Frame: Baseline and End of Treatment (6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CCNMES | Cyclic NMES
Number analyzed (Participants) | 2 | 3
units on a scale | 1 (1.4) | 1.7 (2.9)

2. Secondary Outcome: Change in 10-Meter Walk Test
Description: Time to walk 10 m was measured using a stop-watch. For each individual, the time to walk 10 m prior to treatment was subtracted from the time to walk 10 m at end of the 6-week treatment. Then for each treatment group, these changes in time were averaged.
Time Frame: Baseline and End of Treatment (6 weeks)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | CCNMES | Cyclic NMES
Number analyzed (Participants) | 2 | 3
seconds | 2.2 (7.6) | 0.5 (1.7)

3. Secondary Outcome: Change in Ankle Movement Tracking Error at End of Treatment
Description: Ankle dorsiflexion angle was measured continuously using an electrogoniometer. The subject was seated in front of a computer screen which displayed a 30-sec long sine-wave trace scrolling right to left across the screen. The peak to peak amplitude of the sine wave was set equal to the participant's achievable active range of ankle movement and put on a scale of 0 to 100. Three 30-sec trials were run in which the participant's task was to trace the sine wave by moving their paretic ankle. Error was calculated as the average vertical distance between the sine wave and the ankle angle. The lowest error across three trials was taken as the error for that time point.
  Lower errors are considered to be better outcomes.
  For each participant, the error prior to treatment was subtracted from the error at end of the 6-week treatment. Then for each treatment group, these change scores were averaged. A negative change in error scores is considered an improvement.
Time Frame: Baseline and End of Treatment (6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CCNMES | Cyclic NMES
Number analyzed (Participants) | 2 | 3
units on a scale | -2.6 (4.6) | 4.0 (3.4)

4. Secondary Outcome: Change in Modified Emory Functional Ambulation Profile (MEFAP) at End of Treatment
Description: The MEFAP is a measure of functional ambulation, measuring the time to ambulate through 5 common environmental terrains: 1) 5-meter walk on a hard floor, 2) 5-meter walk on a carpeted floor, 3) rise from a chair, 3-meter walk, return to seated position, 4) standardized obstacle course (bricks to step over), 5) stair ascent and descent. The five times subscores were added to derive a total time.
  Lower times are considered to be a better outcome.
  For each individual, the MEFAP completion time prior to treatment was subtracted from the MEFAP completion time at end of the 6-week treatment. Then for each treatment group, these change values were averaged.
Time Frame: Baseline and End of Treatment (6 weeks)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | CCNMES | Cyclic NMES
Number analyzed (Participants) | 2 | 3
seconds | 2.5 (9.6) | -16.1 (11.1)

ADVERSE EVENTS:
Arm/Group | CCNMES | Cyclic NMES
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes